CLINICAL TRIAL: NCT06258538
Title: Effects of Circuit Training Combining Different Types of Distal Robot-assisted and Task-oriented Therapy on Motor Control, Motor and Daily Functions, and Quality of Life After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202301367B0
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-02

CONDITIONS: Stroke Patients
Keywords: Stroke rehabilitation; distal upper extremity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- distal robot-assisted and task-oriented therapy (Experimental): Participants in the Circuit group received interventions for 20-min exoskeleton(EXO) and 20-min end-effector(EE) robot-assisted therapy, followed by 20-min uni- and 20-min bi- task-oriented therapy/session, 3 sessions/week for 6 consecutive weeks.
  Interventions: Device: Robots can aid in distal UE rehabilitation through exoskeleton (EXO); Device: End-effector robot-assisted therapy (EE); Behavioral: Unilateral task-oriented therapy; Behavioral: Bilateral task-oriented therapy
- distal robot-assisted therapy alone (Experimental): Participants in the Robot group received interventions for 40-min exoskeleton(EXO) and 40-min end-effector(EE) robot-assisted therapy/session, 3 sessions/week for 6 consecutive weeks.
  Interventions: Device: Robots can aid in distal UE rehabilitation through exoskeleton (EXO); Device: End-effector robot-assisted therapy (EE)
- task-oriented therapy alone (Active Comparator): Participants in the task-oriented therapy(TOT) group received interventions for 40-min uni- and 40-min bi- task-oriented therapy/session, 3 sessions/week for 6 consecutive weeks.
  Interventions: Behavioral: Unilateral task-oriented therapy; Behavioral: Bilateral task-oriented therapy

INTERVENTIONS:
Device: Robots can aid in distal UE rehabilitation through exoskeleton (EXO) — Exoskeleton robot-assisted therapy Each EXO robot-assisted therapy session consists of continuous passive motion (30 percent of duration), active-assisted training (30 percent of duration), and interactive training (40 percent of duration) using the Hand of Hope (HOH) robotic hand system . HOH is an exoskeleton type of robot that is worn on the dorsal side of the impaired hand with 2 surface EMG sensors attached to the extensor digitorum and flexor digitorum superficialis.
  Arms: distal robot-assisted and task-oriented therapy; distal robot-assisted therapy alone
Device: End-effector robot-assisted therapy (EE) — Each EE robot-assisted therapy session consists of continuous passive motion (30 percent of duration), active-assisted training (30 percent of duration), and interactive training (40 percent of duration) using the Amadeo robotic system. Amadeo is an end-effector robot with 5 finger slides, which are attached to the fingertips and the thumb via magnetic finger pads. The integrated sensor for each finger allows the robot system to provide patients with real-time visual feedback of finger strengths and range of motion
  Arms: distal robot-assisted and task-oriented therapy; distal robot-assisted therapy alone
Behavioral: Unilateral task-oriented therapy — The therapy will focus on task-oriented therapy with the affected UE and the training tasks involve proximal or distal UE movement, such as ringing a bell, picking up coins, grasping and releasing various cups, and other functional movements involved in daily activities. The level of challenge will be adapted according to patient ability and improvement during training.
  Arms: distal robot-assisted and task-oriented therapy; task-oriented therapy alone
Behavioral: Bilateral task-oriented therapy — The functional training tasks emphasize UE movements (gross or fine motor tasks) involved in daily activities but focus on both UEs moving synchronously, such as opening 2 closet doors, grasping and releasing 2 towels, wiping the table with 2 hands, and so on. The activities can also be graded in terms of difficulty and task requirements, according to the impairment level and the progression of the UE of each participant.
  Arms: distal robot-assisted and task-oriented therapy; task-oriented therapy alone

SUMMARY:
This study proposes a novel stroke rehabilitation approach for upper extremity training by firstly combining different types of distal robot-assisted and task-oriented therapy in a circuit training program. The program could enhance UE functions, improving daily function, decrease caregiver burden and lower medical expenses associated with long-term care. Professionals can use these findings to promote the application of clinically empirical research and better understand the effects and mechanisms of circuit training.

ELIGIBILITY:
Inclusion Criteria:

1. unilateral stroke ≥ 3 months onset
2. Fugl-Meyer Assessment for Upper Extremity (FMA-UE) score between 18 to 56, indicating different levels of motor impairments ;
3. without excessive spasticity in any of the UE joint (modified Ashworth scale ≤3 in proximal joints and modified Ashworth scale ≤2 in distal joints);
4. Mini Mental State Exam (MMSE) score > 24, indicating no serious cognitive impairment;
5. between the ages of 20 and 75 years -

Exclusion Criteria:

1. histories of other neurological diseases such as dementia, Parkinson's disease, and peripheral polyneuropathy;
2. difficulties in following and understanding instructions such as global aphasia;
3. enroll in other rehabilitation or drug studies simultaneously;
4. receiving Botulinum toxin injections within 3 months. -

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The MMSE is a 30-point questionnaire that is the most commonly used brief screening tool for detecting cognitive impairment. Higher values represent better cognitive functioning. The MMSE has good psychometric properties for identifying cognitive impairment
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The upper-extremity subscale of FMA will be used to assess sensorimotor impairment. The FMA-UE includes 33 items assessing movements, reflexes, and coordination of upper limbs. Each item is measured on a 3-point ordinal scale and the total score ranges from 0 to 66 . A higher score indicates better motor function.
  The reliability and validity of the Fugl-Meyer Assessment are well established
Modified Ashworth scale of muscle spasticity (MAS) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The MAS is a 6-point ordinal scale assessing muscle tone, where higher scores represent spasticity. The MAS scores of proximal and distal arm muscles will be examined. The MAS has good validity and reliability
Grip and pinch strength | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The Jamar dynamometer is a standard, accurate, adjustable-handle tool specifically for measuring grip and pinch strength .
  Participants are asked to perform tasks under unilateral and bilateral conditions. In the unilateral condition, participants are asked to exert only with their paretic hands; in the bilateral condition, participants are asked to exert with both hands. Three trials will be taken at each assessment, and the average of three trials will be documented.
Medical Research Council scale (MRC) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The MRC is an ordinal scale assessing muscle strength. The scoring for each muscle ranges from 0 to 5, with a higher score indicates greater muscle strength. The reliability of MRC was good to excellent in stroke patients
Revised Nottingham Sensory Assessment (rNSA) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The rNSA will be used to evaluate changes in sensation. It equips with various sensory modalities to assess tactile sensation, proprioception, and stereognosis of different segments of the body . Scoring of rNSA is based on a 3-point ordinal scale (0-2), with a lower score suggesting greater sensory impairment. The psychometric properties have been established in stroke patients
Wolf Motor Function Test (WMFT) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The WMFT assesses upper extremity motor ability by measuring the performance time (WMFT-Time) and functional ability rating scale (WMFT-FAS) in required task. Participants were timed and rated by using a 6-point ordinal scale. The WMFT is valid and reliable on assessing motor function in stroke patients
Motor Activity Log (MAL) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The MAL falls within the activity and participation domains of ICF framework. It is a semi-structured interview for stroke patients to assess the amount of use (MAL-AOU) and quality of movement (MAL-QOM) of their affected arm and hand during 30 activities of daily living. The score of each activity ranges from 0 to 5, and higher scores represent more frequently used or higher quality of movement. The MAL has good validity, reliability, and responsiveness in patients with stroke
Nottingham Extended Activities of Daily Living Scale (NEADL): | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The NEADL is a measure of independence in 4 areas of daily life, including mobility, kitchen, domestic, and leisure activities. It includes 22 items, and each item is measured on a 4-point scale. The total score ranges from 0 to 66 and a higher score indicates better daily functional ability. The psychometric properties of the NEADL have been well established.
Stroke Impact Scale Version 3.0 (SIS 3.0) | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The SIS 3.0 is a stroke-specific health-related quality of life instrument. It consists of 59 items grouped into 8 domains (strength, hand function, ADL/instrumental ADL, mobility, communication, emotion, memory and thinking, and participation/role function). The participants will be asked to rate each item on a 5-point Likert scale for the perceived difficulty in completing the task. An extra question will be asked to evaluate the participant's self-perceived overall recovery from stroke. The SIS 3.0 has satisfactory psychometric properties in stroke patients
The stroke self-efficacy questionnaires (SSEQ): | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The SSEQ measures an individual's confidence in relation to functional performance and self-management after stroke. It includes 13 items, and each item is rated on a 10-point scale from 0 (not at all confident) to 10 (very confident). The reliability and validity of the SSEQ are well established
Daily Living Self-Efficacy Scale (DLSES): | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The DLSES measures self-efficacy of daily functioning, including psychosocial functioning and activities of daily living. The scale consists of 12 items, and each item is measured on a 100-point scale with 10-unit intervals (0 = cannot do at all, 100 = highly certain can do). A higher score indicates a higher level of self-efficacy. The DLSES is a psychometrically sound measure of self-efficacy in stroke survivors
Functional Abilities Confidence Scale (FACS): | baseline , after the completion of the 18-session intervention , and 3 month after intervention
  The FACS measures the degree of selfefficacy and confidence when the participants perform various movements and postures. It consists of 15 questions scoring from 0% (not confidence at all) to 100% (fully confidence). A higher score indicates higher confidence in performing the movements. The psychometric properties are good

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, Taiwan